CLINICAL TRIAL: NCT05375773
Title: A Single-center, Open-label, Randomized Controlled Trial to Evaluate the Efficacy of Sino-nasal and Mouth Cavity Rinse With an Iodine-based Solution in Reducing Viral Load in Asymptomatic Coronavirus Diseases (COVID-19)
Brief Title: Povidone Iodine Nasal Irrigation and Gargling to Reduce Viral Load in Asymptomatic Patients With COVID-19
Acronym: SMART-CORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, WU Beiwen, clinical nursing professor, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: xmq21966
Record Dates: First submitted 2022-05-15; First posted 2022-05-17 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: 2019 Novel Coronavirus Infection
Keywords: Povidone-Iodine; Nasal Lavage and gargling
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the Control group accept standard treatment for the management of their symptoms according to the diagnosis and treatment for novel coronavirus pneumonia (Trial Nine Edition).
- PVP-I Nasal Irrigation and gargling (Experimental): Participants in the intervention arm will be required to perform Nasal Irrigation and gargling 4 times daily. They will also accept standard treatment for the management of their symptoms according to the diagnosis and treatment for novel coronavirus pneumonia (Trial Nine Edition).
  Interventions: Other: PVP-I Nasal Irrigation and gargling

INTERVENTIONS:
Other: PVP-I Nasal Irrigation and gargling — The solution is prepared by the researcher, which contains 0.5% PVP-I and 2.27% hypertonic saline
  Arms: PVP-I Nasal Irrigation and gargling

SUMMARY:
The emergence of a novel coronavirus(SARS-CoV-2) in late 2019 has resulted in a global epidemic of the infectious condition COVID-19. Since March 2022, the Omicron mutant has caused widespread transmission in Shanghai, China, and is characterized by the majority of asymptomatic patients. Although showing no obvious symptoms, the asymptomatic patients have high transmissibility because of high viral loads in their oropharynx and nasopharynx. Therefore，this study puts forwards the hypothesis that local flushing treatment in the sino-nasal and mouth cavity can reduce the viral load to reduce their transmissibility.

Nasal Irrigation and gargling is a safe and commonly used mechanism to treat a variety of sinonasal diseases including sinusitis, rhinitis, and upper respiratory tract infections. Povidone-iodine(PVP-I) is a water-soluble complex of povidone, a carrier molecule, and iodine, which has powerful microbicidal activity. Also, recent evidence of in-vitro virucidal action of povidone-iodine in Severe Acute Respiratory Syndrome-Coronavirus 2 (SARS CoV-2) has been supported.

Therefore, the study is designed to assess the virucidal effect of nasal irrigation and gargling with PVP-I against SARS-CoV-2 located in the throat. The hypothesis was that the treatment would be effective in improving the negative conversion rate of SARS-CoV-2 nucleic acid on day 10.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate if using nasal irrigation and gargling with PVP-I and hypertonic saline solution, can improve the negative conversion rate of SARS-CoV-2 nucleic acid on day 10 and reduce the incidence rate and severity of symptoms associated with COVID-19.

The study is a prospective, single-center, open-label, randomized controlled trial. The subjects who met the inclusion criteria were stratified according to gender, and randomly divided into control group and experimental group. Both groups were treated according to the diagnosis and treatment for novel coronavirus pneumonia (Trial Nine Edition). Of them, the control group is as blank control, and the experimental group was rinsed with PVP-I containing hypertonic lotion prepared by 0.9% Normal saline（NS）, 10% sodium chloride（NaCl）, and povidone-iodine（PVP-I） gargle four times a day.

The participants in the control group and the experimental group will be required to fill in a daily record and report the main complaint of discomfort. The subjects in the experimental group are also asked to record the implementation of oral and nasal flushing every day.

The researchers are going to record the test results of novel coronavirus nucleic acid samples from the nasopharynx of all subjects in the control group and the experimental group every day.

ELIGIBILITY:
Inclusion Criteria:

* Patients nucleic acid testing positive for COVID-19.
* Diagnose as asymptomatic patients infected by COVID-19, and receive medical observation at a Fang Chang Hospital.
* Be able to understand this study, willing to participate in, and sign the informed consent form.
* Commit to follow the research procedures and cooperate in the implementation of the whole process research.
* Can communicate with researchers through smart phones.

Exclusion Criteria:

* The nucleic acid test result of novel coronavirus has always been negative after entering the Fang Chang Hospital.
* patients who have history of nasal surgery, or current use of nasal saline irrigation or other intranasal medications.
* Patients with thyroid diseases , respiratory diseases or other serious basic diseases.
* Allergy to iodine.
* Participation in another prospective COVID related research project(clinical trial).
* Pregnancy or lactation
* Patients with immune deficiency (such as patients with malignant tumors, organ or bone marrow transplantation, patients with AIDS, and those taking immunosuppressive drugs within 3 months before screening).
* Other patients considered unsuitable by the investigator to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-04-16 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
negative conversion rate | the 10th day after entering the Fang Chang Hospital
  On the 10th day after entering the Fang Chang Hospital, the negative conversion rate of novel coronavirus nucleic acid detected by nasopharyngeal sampling. the "turning negative" is defined as the person whose nucleic acid detection is negative for two times after an interval of more than 24 hours according to the diagnosis and treatment for novel coronavirus pneumonia (Trial Nine Edition).

SECONDARY OUTCOMES:
negative conversion rate | the 5th 、7th and 14th day after entering the Fang Chang Hospital
  the negative conversion rate of novel coronavirus nucleic acid detected by nasopharyngeal sampling
the length of time for patient s when nucleic acid result turns to be negative | 1-14 days or until the nucleic acid result is negative
  Number of days
Intraoral viral load | 10th day of using Nasal Irrigation and gargling
  Intraoral viral load as deciphered by Reverse transcription polymerase chain reaction (RT-PCR) testing
Number of participants reporting side effects of nasal irrigation | 1-14 days or until the participant reports that they are well
  Number of participants in intervention arm reporting side effects
Self-reported clinical discomfort | 1-14 days or until the participant reports that they are well
  Number of participants reported, including headache, cough, runny nose, chest pain, fever, muscle soreness / fatigue, diarrhea / nausea / vomiting, loss of taste / smell and other symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital,Shanghai Jiaotong University school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zou L, Ruan F, Huang M, Liang L, Huang H, Hong Z, Yu J, Kang M, Song Y, Xia J, Guo Q, Song T, He J, Yen HL, Peiris M, Wu J. SARS-CoV-2 Viral Load in Upper Respiratory Specimens of Infected Patients. N Engl J Med. 2020 Mar 19;382(12):1177-1179. doi: 10.1056/NEJMc2001737. Epub 2020 Feb 19. No abstract available. PMID 32074444
- [Background] Koksal T, Cizmeci MN, Bozkaya D, Kanburoglu MK, Sahin S, Tas T, Yuksel CN, Tatli MM. Comparison between the use of saline and seawater for nasal obstruction in children under 2 years of age with acute upper respiratory infection. Turk J Med Sci. 2016 Jun 23;46(4):1004-13. doi: 10.3906/sag-1507-18. PMID 27513397
- [Background] Slapak I, Skoupa J, Strnad P, Hornik P. Efficacy of isotonic nasal wash (seawater) in the treatment and prevention of rhinitis in children. Arch Otolaryngol Head Neck Surg. 2008 Jan;134(1):67-74. doi: 10.1001/archoto.2007.19. PMID 18209140
- [Background] Ramalingam S, Graham C, Dove J, Morrice L, Sheikh A. A pilot, open labelled, randomised controlled trial of hypertonic saline nasal irrigation and gargling for the common cold. Sci Rep. 2019 Jan 31;9(1):1015. doi: 10.1038/s41598-018-37703-3. PMID 30705369
- [Background] Ramalingam S, Cai B, Wong J, Twomey M, Chen R, Fu RM, Boote T, McCaughan H, Griffiths SJ, Haas JG. Antiviral innate immune response in non-myeloid cells is augmented by chloride ions via an increase in intracellular hypochlorous acid levels. Sci Rep. 2018 Sep 11;8(1):13630. doi: 10.1038/s41598-018-31936-y. PMID 30206371
- [Background] Vogt PM, Hauser J, Mueller S, Bosse B, Hopp M. Efficacy of Conventional and Liposomal Povidone-Iodine in Infected Mesh Skin Grafts: An Exploratory Study. Infect Dis Ther. 2017 Dec;6(4):545-555. doi: 10.1007/s40121-017-0172-z. Epub 2017 Oct 10. PMID 29019097
- [Background] Eggers M, Koburger-Janssen T, Eickmann M, Zorn J. In Vitro Bactericidal and Virucidal Efficacy of Povidone-Iodine Gargle/Mouthwash Against Respiratory and Oral Tract Pathogens. Infect Dis Ther. 2018 Jun;7(2):249-259. doi: 10.1007/s40121-018-0200-7. Epub 2018 Apr 9. PMID 29633177
- [Background] Kariwa H, Fujii N, Takashima I. Inactivation of SARS coronavirus by means of povidone-iodine, physical conditions and chemical reagents. Dermatology. 2006;212 Suppl 1(Suppl 1):119-23. doi: 10.1159/000089211. PMID 16490989
- [Background] Eggers M, Eickmann M, Zorn J. Rapid and Effective Virucidal Activity of Povidone-Iodine Products Against Middle East Respiratory Syndrome Coronavirus (MERS-CoV) and Modified Vaccinia Virus Ankara (MVA). Infect Dis Ther. 2015 Dec;4(4):491-501. doi: 10.1007/s40121-015-0091-9. Epub 2015 Sep 28. PMID 26416214
- [Background] Anderson DE, Sivalingam V, Kang AEZ, Ananthanarayanan A, Arumugam H, Jenkins TM, Hadjiat Y, Eggers M. Povidone-Iodine Demonstrates Rapid In Vitro Virucidal Activity Against SARS-CoV-2, The Virus Causing COVID-19 Disease. Infect Dis Ther. 2020 Sep;9(3):669-675. doi: 10.1007/s40121-020-00316-3. Epub 2020 Jul 8. PMID 32643111
- [Background] Arefin MK, Rumi SKNF, Uddin AKMN, Banu SS, Khan M, Kaiser A, Chowdhury JA, Khan MAS, Hasan MJ. Virucidal effect of povidone iodine on COVID-19 in the nasopharynx: an open-label randomized clinical trial. Indian J Otolaryngol Head Neck Surg. 2022 Oct;74(Suppl 2):2963-2967. doi: 10.1007/s12070-021-02616-7. Epub 2021 May 18. PMID 34026595